CLINICAL TRIAL: NCT04409925
Title: Phase I Pilot Study Investigating the Safety and Feasibility of Inhaled rhDNase1 and Its Impact on Neutrophil Extracellular Traps (NETs) in Non-Ventilated COVID-19 Infected Patients
Brief Title: DISmantling COvid iNduced Neutrophil ExtraCellular Traps (DISCONNECT-1)
Acronym: DISCONNECT-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); Hoffmann-La Roche (Industry); Exactis Innovation (Other)
Responsible Party: Principal Investigator, Jonathan Spicer, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DISCONNECT-1
Record Dates: First submitted 2020-05-13; First posted 2020-06-01 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: COVID-19 Infection
Keywords: Neutrophil Extracellular Traps; NETs; Neutrophils; rhDNase1
MeSH Terms: conditions — COVID-19 | interventions — dornase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- rhDNase1 (Pulmozyme, Roche/Genentech) (Experimental): Single Arm: rhDNase1 (Pulmozyme, Roche/Genentech) 2.5 mg inhaled nebulisations BID, for a maximum of 14 consecutive days.
  Interventions: Drug: rhDNase I

INTERVENTIONS:
Drug: rhDNase I — Inhaled nebulisations
  Other Names: Pulmozyme

SUMMARY:
This is a pilot study to investigate the safety and feasibility of rhDNase1 and its impact on neutrophil extracellular traps (NETs) in COVID-19 infected patients.

DETAILED DESCRIPTION:
It has been reported that elevated numbers of neutrophils (PMNs) in the blood predicts poor outcomes and severity in patients with COVID-19 infections. Acute inflammation results in formation of neutrophil extracellular traps (NETs) by PMNs and NK cells. Pre-clinical studies showed that NETs are critically involved in the pathophysiology of ARDS and increased capacity of PMNs to form NETs was shown to correlated with increased severity and mortality in patients with ARDS after community-acquired pneumonia. In early reports, patients with severe COVID-19 infections were also found to have radiological and clinical findings of Acute Respiratory Distress Syndrome (ARDS). NETs can be degraded by DNase1 for which there is a human recombinant equivalent rhDNase1.

This study proposes:

1. to evaluate the safety and feasibility of inhaled rhDNase1 in severely ill COVID-19 patients requiring admission;
2. to evaluate the impact of rhDNase1 in limiting progression of disease and COVID-19 related complications in these patients;
3. and to investigate NETs as possible therapeutic targets in severe COVID-19 patients by quantifying levels of circulating NETs in the blood and sputum and correlating these with oxygen requirements, need for mechanical ventilation, duration of mechanical ventilation, radiological progression of ARDS, secondary bacterial infections (pneumonia, bacteremia and other), renal dysfunction, duration of ICU admission, and time to discharge or mortality.

ELIGIBILITY:
Inclusion criteria

1. Verbal informed consent by patient (or legal representative), done in the presence of an impartial witness. The consent is signed by the Principal Investigator (or Co-Investigator) and the impartial witness.
2. Participants who are at least 18 years of age on the day of consenting to the informed consent
3. COVID-19 (SARS-CoV2) positive test by nasopharyngeal swab
4. Admitted to the ICU in negative pressure rooms
5. Mild to severe respiratory illness (defined as requiring admission* and/or supplemental oxygen), not intubated or on mechanical ventilation at screening and enrolment.

   * Admission respiratory criteria (1 of the following):

     1. Dyspnea at rest or during minimal activity (sitting, talking, coughing, swallowing);
     2. Respiratory rate > 22/minute;
     3. PaO2 < 65mmHg or oxygen saturation < 90% or PaO2/FiO2 ratio of less than 300
     4. Infiltrate on CXR (or worsening CXR, if baseline CXR at admission was already abnormal)
   * Mild disease with hospitalization:

     * No oxygen therapy;
     * Oxygen by mask or nasal prongs.
   * Severe disease with hospitalization (requiring greater than 40% oxygen):

     * Oxygen by non-invasive ventilation or high flow oxygen/Optiflow.

Exclusion criteria:

1. Patients requiring mechanical ventilation at screening
2. Previous or current treatment with rhDNase1
3. Ongoing experimental treatment with other inhaled therapies through COVID-19-related clinical trials
4. Known hypersensitivity to NET inhibitor or recombinant protein products
5. Known hypersensitivity to Chinese Hamster Ovary cell products or any component of the product
6. Known history of immunodeficiency, HBV, HCV, HIV (Note: No HBV, HCV or HIV testing is required unless mandated by local health authority)
7. Known history of immunosuppressive disorders, such as primary/secondary immunodeficiencies, lymphoproliferative diseases
8. Active pregnancy at any stage or lactation
9. Patients deemed incapable and/or incompetent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-25 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Safety of inhaled rhDNase1 in non-ventilated COVID-19 patients by reporting of adverse events | 9 months
  Rate of all adverse events, rate of serious adverse events, rate of grade 3/4/5 adverse events, rate of drug-related adverse events.

SECONDARY OUTCOMES:
Time to first study participant enrolment | Up to 2 weeks
  Time elapsed between the study opening date and the first patient enrolment date.
Enrolment rate | Up to 9 months
  Number of patients enrolled per week following the start of the study.
Eligible patient consent rate | Up to 9 months
  Number of patients meeting eligibility through inclusion and exclusion criteria that are consented and enrolled into the study, as compared to the total number of patients meeting criteria (enrolled and non-enrolled).
Completeness of drug delivery | Up to 9 months
  Percentage of doses missed compared to completed, including reasons for missed doses, per patient.
Completeness of study-specific tests or procedures | Up to 9 months
  Percentage of tests or procedures missed compared to completed, per patient.
Completeness of data collection | Up to 9 months
  Percentage of missed data compared to completed data, per patient.
Hypoxia rate | Up to 9 months
  Extent of hypoxia rate is defined as the number of patients requiring supplemental oxygen, categorized by type of oxygen requirement.
Supplemental oxygen requirement type | Up to 9 months
  Type of oxygen in FiO2 requirements needed by each patient in the study, if applicable.
Progression to mechanical ventilation rate | Up to 9 months
  Number of patients progressing to requiring intubation and mechanical ventilation.
Duration of mechanical ventilation | Up to 9 months
  Duration in days, for patients requiring intubation and mechanical ventilation, if applicable.
Radiological progression | Up to 9 months
  Number of patients who show progression on imaging suggestive of ARDS such as bilateral lung involvement, as reviewed by study's thoracic radiologist.
Renal dysfunction rate | Up to 9 months
  Number of patients with renal dysfunction, classified by stage (1, 2 or 3).
Renal dysfunction extent | Up to 9 months
  Extent of change in creatinine from baseline.
Secondary bacterial infections rate | Up to 9 months
  Number of patients contracting secondary bacterial infections (pneumonia, bacteremia and other).
Duration of ICU admission | Up to 9 months
  In days, length of stay in the ICU.
Time to hospital discharge or in-hospital mortality | Up to 9 months
  Time elapsed between enrolment into the study (at admission), and endpoint (discharge from ICU or in-hospital mortality).

OTHER OUTCOMES:
Exploratory: NET quantification in blood, correlated to COVID-19 disease severity and complications. | Up to 9 months
Exploratory: Blood clotting and fibrinolysis assays, correlated to COVID-19 disease severity and complications. | Up to 9 months
Exploratory: Cytokine profile alterations in blood, correlated to COVID-19 disease severity and complications | Up to 9 months
Exploratory: Neutrophil RNA sequencing in blood, correlated to COVID-19 disease severity and complications | Up to 9 months
Length of PCR positivity | Up to 9 months
  Defined as number of days between first positive PCR test and last positive PCR test, usually done by nasopharyngeal swabs. Tests will be performed as mandated by standard of care only.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Spicer, MD, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Canada (2):
  - Hamilton General Hospital, Hamilton Health Sciences, Hamilton, Ontario
  - McGill University Health Centre, Montreal, Quebec